CLINICAL TRIAL: NCT04802434
Title: Randomized Controlled Trial of Strengthening Skills, A Multi-Component Behavioral Intervention to Increase Functional Independence During Aging in Autism Spectrum Disorder
Brief Title: Strengthening Skills Behavioral Intervention for Adults With Autism Spectrum Disorder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Southwest Autism Research & Resource Center (Other)
Collaborators: Arizona State University (Other); Mayo Clinic (Other)
Responsible Party: Principal Investigator, Nicole Matthews, Ph.D., Director of Research, Southwest Autism Research & Resource Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 00011585; W81XWH-20-1-0171 (Other Grant/Funding Number: Department of Defense CDMRP)
Record Dates: First submitted 2021-03-12; First posted 2021-03-17 (Actual); Last update posted 2023-11-22 (Actual); Status verified 2023-11

CONDITIONS: Autism Spectrum Disorder
MeSH Terms: conditions — Autism Spectrum Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Strengthening Skills Program (Experimental): Adults with ASD and their study partners (i.e., spouse, parent, other family member, or friend) will attend weekly 3 hour meetings for 16 weeks, during which, behavioral intervention strategies will be used to teach cognitive compensation and mindfulness-based emotion regulation skills. Strategies from the PEERS Social Skills Program will also be taught. Participants will be assigned homework assignments each week to practice skills they are learning in a real-world setting.
  Interventions: Behavioral: Strengthening Skills Program; Behavioral: PEERS Social Skills Program
- PEERS Social Skills Program (Active Comparator): Adults with ASD and their study partners (i.e., spouse, parent, other family member or friend) will attend weekly 1.5 hour meetings for 16 weeks, during which, behavioral intervention strategies will be used to teach skills for improving social relationships and handling social rejection. Participants will be assigned homework assignments each week to practice skills they are learning in a real-world setting.
  Interventions: Behavioral: PEERS Social Skills Program
- Delayed Treatment Control Group (No Intervention): Participants in the delayed treatment control group will participate in a 10-month wait period, during which they will complete data collection procedures at three time points (Baseline, Post, and 6-month follow-up).

INTERVENTIONS:
Behavioral: Strengthening Skills Program — The Strengthening Skills Program is a new, multi-component intervention. It includes three components: (1) Forming habits to compensate for the difficulties many adults with ASD have with thinking flexibly, planning, and time management. It will emphasize habit-forming behaviors to compensate for weaknesses in functional skills by training on practical techniques; (2) Content from the PEERS Social Skills program to target social challenges, and (3) strategies derived from Mindfulness Based Stress Reduction to target emotion regulation.
  Arms: Strengthening Skills Program
Behavioral: PEERS Social Skills Program — PEERS® is a well-established social communication training program, initially developed for adolescents, and more recently extended to young adults with ASD. Program content will be adapted slightly so as to be appropriate for older adults.
  Arms: PEERS Social Skills Program; Strengthening Skills Program

SUMMARY:
The purpose of this study is to examine changes in adaptive functioning, quality of life, and prospective memory among adults with ASD (Autism Spectrum Disorder) who complete Strengthening Skills, a multi-faceted, behavioral intervention that combines the PEERS Social Skills program with cognitive compensation training, mindfulness-based emotional regulation, and support group components. Participants and their study partners (e.g., spouse, parent, friend) will be randomly assigned to one of three groups: Strengthening Skills, PEERS only, or a delayed treatment control group. The Strengthening Skills group will meet weekly for 3 hours for 16 weeks and will learn strategies for gaining and maintaining independence and emotion regulation. Participants will also learn strategies from the PEERS Social Skills Program. The PEERS only group will meet weekly for 1.5 hours for 16 weeks and will only learn strategies from the PEERS Social Skills Program. The delayed treatment control group will participant in data collection at four time points over a 10-month wait period, after which, they will be enrolled into the Strengthening Skills Program. Behavioral self-report data will be collected and a prospective memory assessment will be conducted before and after participation in the 16-week programs. Behavioral self-report data will also be collected at remote 3- and 6-month follow-up visits.

ELIGIBILITY:
Inclusion Criteria:

* Meets criteria for autism or autism spectrum on a gold-standard diagnostic assessment (Autism Diagnostic Observation Schedule-2)
* Must have a study partner (e.g., parent, spouse, sibling, friend) willing and able to complete questionnaires at all four time points
* Must be willing to be randomized to a treatment or delayed treatment control group
* Must be able to attend at least 14 of the 16 weekly intervention sessions
* English speaking: Participants must be English-speaking because the screening and behavioral measures are in English (including the intelligence estimate), as well as the intervention content

Exclusion Criteria:

* Non-verbal participants will be excluded to ensure test compliance and increase sample homogeneity.
* Participants with IQ (intelligence quotient) scores lower than 70 will be excluded because the interventions were developed for individuals without intellectual disability.

Ages: 21 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2021-04-01 (Actual); Primary Completion 2023-04-30 (Actual); Study Completion 2023-04-30 (Actual)

PRIMARY OUTCOMES:
Mean Change from Baseline in Adaptive Functioning on the Adaptive Behavior Assessment System, Third Edition (ABAS-3) | Post-Intervention (16 weeks); 3-month follow-up; 6-month follow-up
  The ABAS-3 Adult Form is a self and other-report questionnaire designed specifically for adult participants (ages 16 to 89), which yields standard scores (Mean = 100, Standard Deviation = 15) in three adaptive domains (i.e., Conceptual, Social, and Practical) and a General Adaptive Composite (GAC). Scores range from 40 to 120 with higher scores indicating better adaptive functioning.
Mean Change from Baseline in Self-reported Quality of Life on the World Health Organization's Brief Quality of Life assessment (WHOQOL-BREF) | Post-Intervention (16 weeks); 3-month follow-up; 6-month follow-up
  The WHOQOL-BREF is an abbreviated version of the World Health Organization's Quality of Life assessment (WHOQOL-100). 26-item self-report questionnaire that yields an Overall Quality of Life and General Health score and four quality of life domain scores: physical health, psychological, social relationships, and environment. Scores range from 0 to 100 on all domains, with higher scores indicating better quality of life.

SECONDARY OUTCOMES:
Mean Change from Baseline in Prospective Memory on the Royal Prince Alfred Prospective Memory Test | Post-Intervention (16 weeks)
  4-item behavioral measure of prospective memory. Each item has a maximum score of three points, with a total possible score of 12 points. Scores range from 0 to 12, with higher scores indicating better prospective memory.

CONTACTS AND LOCATIONS:
Overall Officials: Nicole L Matthews, Ph.D., Principal Investigator — Southwest Autism Research & Resource Center; Brittany B Braden, Ph.D., Principal Investigator — Arizona State University
Locations (1):
- Arizona State University, Tempe, Arizona, United States

IPD SHARING:
Plan to Share IPD: Yes
All individual participant data (IPD) that underlie results in a publication will be available upon request to approved researchers.
Supporting Information: Study Protocol
Time Frame: Data will be available upon request starting 6 months after publication and will remain available for 2 years.
Access Criteria: Data requests should be submitted to Dr. Blair Braden at bbbraden@asu.edu and must include study aims and purpose and a detailed analysis plan describing how the data will be used. Requests will be reviewed by Dr. Braden and access to the data will be made available through a secure link to download the requested data.